CLINICAL TRIAL: NCT04664426
Title: Adapted Modified Toronto Clinical Neuropathy Score and Erasmus Polyneuropathy Symptom Score Validated by Quantitative Sensory Testing and Nerve Conduction Studies for Kidney Transplant Recipients
Brief Title: Sensory Neuropathy Scores Validated by Quantitative Sensory Testing and Nerve Conduction Studies for Kidney Transplant Recipients
Acronym: SENS
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Gea Drost, Principal Investigator, University Medical Center Groningen
Other Study IDs: SENS study
Record Dates: First submitted 2020-11-16; First posted 2020-12-11 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Polyneuropathies
Keywords: polyneuropathy; quantitative sensory testing; nerve conduction studies; adapted modified Toronto Clinical Neuropathy Score; renal transplantation; Erasmus Polyneuropathy Symptom Score
MeSH Terms: conditions — Polyneuropathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney transplant recipients: Kidney transplant recipients will undergo examination according to the E-PSS, amTCNS, QST (thermal threshold testing), and NCS (amplitude, velocity and distal latency of measurements at the sural sensory nerve, ulnar sensory nerve, peroneal motor nerve, tibial motor nerve and ulnar motor nerve, soleus H reflex will be measured).

SUMMARY:
Sensory polyneuropathy is one of the most prevalent neurological disorders and a common finding in kidney transplant recipients (KTR). However, prevalence, course and underlying aetiology in this specific patient group remain unexplored. To diagnose sensory polyneuropathy in KTR in clinical practice, a relatively easy and inexpensive method is needed. The Erasmus Polyneuropathy Symptom Score (E-PSS) and the adapted modified Toronto Clinical Neuropathy Score (amTCNS) are such scores. These scores would enable internal medicine physicians to diagnose polyneuropathy in a reliable way without the need of additional examinations. However, a validation of the E-PSS and amTCNS with the golden standard of diagnosing sensory polyneuropathy, which are quantitative sensory testing (QST) and nerve conduction studies (NCS), is needed.

The objective of this observational cross-sectional study is to validate the E-PSS and amTCNS with QST and NCS and to determine reference values of the amTCNS. 200 KTR will be included to take part in one study visit which encompasses neurological examination according to the protocol of the amTCNS, QST and NCS. Prior to the study visit, participants will be asked to answer the E-PSS questionnaire in the home setting.

The main study endpoint is to validate the E-PSS and the amTCNS result with QST and NCS. To reach this endpoint different study parameters will be included which are the result of the E-PSS and amTCNS, results of the QST (thermal threshold testing), and results of the NCS (amplitude, velocity and distal latency of measurements at the sural sensory nerve, ulnar sensory nerve, peroneal motor nerve, tibial motor nerve and ulnar motor nerve, soleus H reflex).

DETAILED DESCRIPTION:
Sensory polyneuropathy is one of the most prevalent neurological disorders. A Dutch study observed an incidence of all types of polyneuropathy of 77 per 100.000 person-years, which increases with age. Besides, previous studies evaluated the impact of polyneuropathy on quality of life in different patient populations and showed that accompanying symptoms affect daily living and influence morbidity and mortality of patients adversely.

We can classify sensory polyneuropathies broadly into either small fibre neuropathies, large fibre neuropathies or mixed small and large fibre neuropathies. In small fibre neuropathies the thinly myelinated A delta and unmyelinated C fibres are affected. Therefore, the transmission of thermal and noxious sensory input is disturbed translating to symptoms of sharp, painful, or burning paraesthesia, sensory loss or numbness, and the inability to discriminate between hot and cold sensation. Disorders affecting the large myelinated A delta fibres lead to an impaired vibration sensation and proprioception. Patients will complain about a combination of symptoms of sensory loss, paraesthesia, and gait imbalance.

Sensory polyneuropathy is a common finding in kidney transplant recipients (KTR), but little is known about prevalence, course, or underlying aetiology in this specific group. It is known that patients are at a high risk to develop polyneuropathy before kidney transplantation due to chronic kidney disease. Therefore, related to the previous state of chronic kidney disease uremic and diabetic polyneuropathy are probable underlying aetiologies in KTR. Furthermore, the use of immunosuppressive medication after transplantation, in particular tacrolimus, may result in polyneuropathic symptoms and signs. These circumstances may explain the high prevalence of polyneuropathy in KTR but in order to gain more understanding, it is necessary to diagnose and stage polyneuropathy in an easy and convenient way in KTR. Furthermore, early diagnosis and treatment of certain types of polyneuropathy can prevent further worsening of neuropathic symptoms and signs, or even reverse the neurologic deficits.

The diagnostic approach to polyneuropathy differs depending on the type of affected nerve fibre and the distribution of nerve damage in the respective type of polyneuropathy. The diagnosis of polyneuropathy is generally based on the presence of distal sensory and sensorimotor symptoms and signs, and loss of function, which is consistent with the clinical picture. Nevertheless, to reveal an underlying large fibre aetiology, nerve conduction studies (NCS) are needed. With the help of NCS, it is possible to categorize polyneuropathy as primary axonal or primary demyelinating. This standard diagnostic test, however, exclusively enables the measurement of large fibres and patients with pure small fibre neuropathies will not show any nerve conduction abnormalities. Hence, quantitative sensory testing (QST) is required to assess the function of small sensory nerve fibres. However, NCS and QST are time-consuming, fairly expensive, and the investigator needs a certain level of expertise. Alternatively, different clinical scores exist that aim to detect and stage polyneuropathy based on symptoms and signs. The Toronto Clinical Neuropathy Score (TCNS) was designed for diabetic sensorimotor polyneuropathy but it was shown that its usefulness extends beyond diabetic polyneuropathy. These results were based on correlations of the TCNS with clinical, electrophysiological and disability parameters in non-diabetic polyneuropathies. The same study confirmed that reliability and accuracy were excellent. Eventually, the TCNS was modified (into the mTCNS) to better capture a scale of simple sensory tests representative of early-stage dysfunction and reflex testing was removed due to its high inter-rater variability. The mTCNS was demonstrated to maintain an acceptable correlation with the precursor score. In the University Medical Center Groningen (UMCG) a large population of KTR is followed within the scope of the TransplantLines cohort study and biobank. For this purpose, the mTCNS was further adapted by omitting testing of temperature sense due to practical reasons (adapted into the amTCNS). The E-PSS was designed to diagnose chronic polyneuropathy and was previously validated in a cohort of patients with chronic idiopathic axonal polyneuropathy.

To be able to study prevalence, course, and underlying aetiology in this specific population of KTR it is crucial to reveal whether the E-PSS and amTCNS correlate with the golden standards of diagnosing polyneuropathy, NCS and QST. In the long term, both clinical scores have great potential to help clinicians from various disciplines without the specific expertise needed for NCS and QST to diagnose polyneuropathy.

In conclusion, the aim of this research proposal is to validate the E-PSS and amTCNS with NCS and QST for a population of KTR.

The primary objective is to validate the Erasmus Polyneuropathy Symptoms Score (E-PSS) and adapted modified Toronto Clinical Neuropathy Score (amTCNS) with QST and NCS.

The secondary objective is to define reference values of the amTCNS dependent on predictors in a healthy subject population. This healthy subject population consists of potential kidney donors that were already seen and examined within the TransplantLines cohort study and biobank prior to this study. These healthy subjects will not undergo QST or NCS.

This research protocol contains a cross-sectional study or can alternatively be described as a validation study. The aim is to examine the validity of the E-PSS and amTCNS, clinical scores that were designed to capture symptoms and signs of sensory polyneuropathy. The E-PSS and amTCNS will be validated with QST and NCS which are defined as golden standards for diagnosing small fibre neuropathies and large fibre neuropathies, respectively.

The aim is to validate the E-PSS and amTCNS for a population of KTR to be able to subsequently identify and follow up on polyneuropathies in this specific population in a more convenient way.

KTR will be recruited retrospectively after their participation in the TransplantLines cohort and biobank study in the UMCG by telephone. Every possible future participant will receive written information concerning this study (aim, design and duration of the study, disadvantages and risks of participation). The subjects will be required to sign the written informed consent form within two weeks if they want to take part in this study. The subjects will be informed that if they give consent for participation in the study they may withdraw consent at any time. This withdrawal of consent may be given to the investigator in oral or written form. After receiving the written informed consent a screening via telephone will be planned to assess whether the potential participant meets the inclusion criteria.

The amTCNS result will be calculated based on a questionnaire and neurological examination. This includes a symptoms score assessing foot pain, numbness, tingling, weakness, ataxia and upper limb symptoms, and a sensory test score including testing of pinprick sensation, light touch, proprioception and vibration sense. QST consists of thermal threshold testing in which the thresholds of warm sensation and cold sensation will be determined following the method of limits and the method of levels. NCS will include testing of the CMAP amplitude and distal motor latency of the tibial, peroneal and ulnar nerve; the SNAP amplitude of the sural and ulnar nerve; nerve conduction velocity and the soleus H-reflex. Participants will be asked to fill in the questionnaire of the E-PSS prior to their study visit via mail.

Prior to this study the amTCNS was already carried out in 200 healthy subjects which were potential kidney donors. Clinical characteristics that function as independent predictors of the amTCNS in a healthy subject population will be determined by means of ordinal logistic regression analyses. The 95th percentile of the amTCNS final score will be calculated to define reference values according to the identified independent predictors. The outcome of the polyneuropathy measures of the current study will be dichotomized as follows: presence of polyneuropathy (both aberrant QST and NCS), presence of small fibre neuropathy (aberrant QST), presence of large fibre neuropathy (aberrant NCS). These outcomes will be opposed to the dichotomous outcome of presence of polyneuropathy according to the reference value of the amTCNS that was previously established in a healthy subject population. Sensitivity, specificity, positive predictive value and negative predictive value will be calculated.

To compare amTCNS cut-off points for diagnosis, the reference values determined in the cohort of healthy subjects without polyneuropathy will be compared with the data in KTR. The accuracy of the amTCNS in KTR will be determined by the area under the receiver operating characteristic curve, with the presence of polyneuropathy as the dichotomous outcome variable and amTCNS as the test. The optimal diagnostic threshold will be identified by the point on the receiver operating characteristic curve closest to the point of perfect discrimination.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 y.o.
* Patient is able to understand the Dutch language and capable to intellectually comprehend questionnaires and physical tests
* Signed and dated informed consent prior to any study-related procedures
* Previous participation in the TransplantLines cohort study and biobank

Exclusion Criteria:

* Patient refusal
* Amputation of lower or upper limb(s), trauma of limbs
* Patients with a pacemaker or ICD
* Use of mind-altering drugs in previous 24 hours
* Metal osteosynthesis after bone fracture (in arms or legs)
* Patients with mononeuropathies in examined nerves
* Patients on dialysis after transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of kidney transplant recipients (KTR).
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
adapted modified Toronto Clinical Neuropathy Score (amTCNS) | First test of the study visit, will be performed once (each study participant has a single study visit), Day 1
  The amTCNS examines signs and symptoms of polyneuropathy. It consists of a questionnaire which explores the presence of neuropathic pain, numbness, tingling, weakness, and loss of sensation leading to ataxia. Secondly, sensory tests will be performed including sensation for pinprick, light touch, proprioception, and vibration. The minimum value is 0 meaning the patient does not show any signs or symptoms of polyneuropathy and the maximum value is 30 meaning the patient presents with severe signs and symptoms of polyneuropathy.
Quantitative sensory testing (QST) | Second test of the study visit, will be performed once (each study participant has a single study visit), Day 1
  Quantitative sensory testing will be performed according to the method of temperature threshold testing. Both the method of limits and the method of levels will be carried out.
Nerve conduction studies (NCS) | Third test of the study visit, will be performed once (each study participant has a single study visit), Day 1
  Sensory nerve action potential (SNAP) amplitude of the sural and ulnar nerve will be recorded and compound muscle action potential (CMAP) amplitude of the tibial, peroneal and ulnar nerve. Furthermore, the soleus Hoffman's reflex will be tested. For all measurements the amplitude (mV), conduction velocity (m/s) and distal latency (ms) of the described nerves will be determined.
Erasmus Polyneuropathy Symptom Score (E-PSS) | Participants will be asked to fill in the six-time questionnaire of the E-PSS prior to their study visit in the home setting via mail.
  The E-PSS consists of a six-item questionnaire taking the presence and frequency of different polyneuropathic symptoms into account.

SECONDARY OUTCOMES:
Muscle strength | Additional testing during the study visit, will be performed once (each study participant has a single study visit), Day 1
  Proximal and distal muscle strength will be tested. Muscle strength testing of the upper extremities will include biceps, triceps and grip strength. In the lower extremities, muscle strength of quadriceps femoris and ankle dorsiflexion will be tested. The testing will be performed using a handheld dynamometer (MicroFET, Draper, UT).
Reflexes | Additional testing during the study visit, will be performed once (each study participant has a single study visit), Day 1
  Biceps brachii, triceps brachii, brachioradialis, quadriceps femoris, triceps surae and plantar reflexes will be tested bilaterally. Reflexes will be described as normal or abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Gea Drost, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be saved under a SENS trial number (STN). The principal investigator has access to the key document (digital). Only members of the study group can access the decoding list. The data collected in the scope of this study will only be used by this study group.

REFERENCES:
- [Background] Abraham A, Alabdali M, Alsulaiman A, Albulaihe H, Breiner A, Katzberg HD, Aljaafari D, Lovblom LE, Bril V. The sensitivity and specificity of the neurological examination in polyneuropathy patients with clinical and electrophysiological correlations. PLoS One. 2017 Mar 1;12(3):e0171597. doi: 10.1371/journal.pone.0171597. eCollection 2017. PMID 28249029
- [Background] Visser NA, Notermans NC, Linssen RS, van den Berg LH, Vrancken AF. Incidence of polyneuropathy in Utrecht, the Netherlands. Neurology. 2015 Jan 20;84(3):259-64. doi: 10.1212/WNL.0000000000001160. Epub 2014 Dec 12. PMID 25503982
- [Background] Senzolo M, Ferronato C, Burra P. Neurologic complications after solid organ transplantation. Transpl Int. 2009 Mar;22(3):269-78. doi: 10.1111/j.1432-2277.2008.00780.x. Epub 2008 Dec 6. PMID 19076332
- [Background] Gwathmey KG. Sensory Polyneuropathies. Continuum (Minneap Minn). 2017 Oct;23(5, Peripheral Nerve and Motor Neuron Disorders):1411-1436. doi: 10.1212/CON.0000000000000518. PMID 28968369
- [Background] Gwathmey KG, Pearson KT. Diagnosis and management of sensory polyneuropathy. BMJ. 2019 May 8;365:l1108. doi: 10.1136/bmj.l1108. PMID 31068323
- [Background] Arnold R, Kwai NC, Krishnan AV. Mechanisms of axonal dysfunction in diabetic and uraemic neuropathies. Clin Neurophysiol. 2013 Nov;124(11):2079-90. doi: 10.1016/j.clinph.2013.04.012. Epub 2013 May 15. PMID 23683523
- [Background] Arnold R, Pianta TJ, Pussell BA, Kirby A, O'Brien K, Sullivan K, Holyday M, Cormack C, Kiernan MC, Krishnan AV. Randomized, Controlled Trial of the Effect of Dietary Potassium Restriction on Nerve Function in CKD. Clin J Am Soc Nephrol. 2017 Oct 6;12(10):1569-1577. doi: 10.2215/CJN.00670117. Epub 2017 Sep 11. PMID 28893921
- [Background] Cengiz N, Adibelli Z, Yakupoglu YK, Turker H. Neurological Complications after Renal Transplantation: A Retrospective Clinical Study. Noro Psikiyatr Ars. 2015 Dec;52(4):331-335. doi: 10.5152/npa.2015.9876. Epub 2015 Dec 1. PMID 28360735
- [Background] Bechstein WO. Neurotoxicity of calcineurin inhibitors: impact and clinical management. Transpl Int. 2000;13(5):313-26. doi: 10.1007/s001470050708. PMID 11052266
- [Background] Arnold R, Pussell BA, Pianta TJ, Lin CS, Kiernan MC, Krishnan AV. Association between calcineurin inhibitor treatment and peripheral nerve dysfunction in renal transplant recipients. Am J Transplant. 2013 Sep;13(9):2426-32. doi: 10.1111/ajt.12324. Epub 2013 Jul 10. PMID 23841745
- [Background] Siao P, Kaku M. A Clinician's Approach to Peripheral Neuropathy. Semin Neurol. 2019 Oct;39(5):519-530. doi: 10.1055/s-0039-1694747. Epub 2019 Oct 22. PMID 31639835
- [Background] Terkelsen AJ, Karlsson P, Lauria G, Freeman R, Finnerup NB, Jensen TS. The diagnostic challenge of small fibre neuropathy: clinical presentations, evaluations, and causes. Lancet Neurol. 2017 Nov;16(11):934-944. doi: 10.1016/S1474-4422(17)30329-0. PMID 29029847
- [Background] Abraham A, Barnett C, Katzberg HD, Lovblom LE, Perkins BA, Bril V. Toronto Clinical Neuropathy Score is valid for a wide spectrum of polyneuropathies. Eur J Neurol. 2018 Mar;25(3):484-490. doi: 10.1111/ene.13533. Epub 2017 Dec 26. PMID 29194856
- [Background] Hanewinckel R, Ikram MA, van Doorn PA. Assessment scales for the diagnosis of polyneuropathy. J Peripher Nerv Syst. 2016 Jun;21(2):61-73. doi: 10.1111/jns.12170. PMID 26968746
- [Background] Bril V, Perkins BA. Validation of the Toronto Clinical Scoring System for diabetic polyneuropathy. Diabetes Care. 2002 Nov;25(11):2048-52. doi: 10.2337/diacare.25.11.2048. PMID 12401755
- [Background] Bril V, Tomioka S, Buchanan RA, Perkins BA; mTCNS Study Group. Reliability and validity of the modified Toronto Clinical Neuropathy Score in diabetic sensorimotor polyneuropathy. Diabet Med. 2009 Mar;26(3):240-6. doi: 10.1111/j.1464-5491.2009.02667.x. PMID 19317818
- [Background] Nolte S, van Londen M, Elting JWJ, de Greef BTA, Kuks JBM, Faber CG, Nolte IM, Groen RJM, Bakker SJL, Groothof D, Lesman-Leegte I, Berger SP, Drost G. Vibration threshold in non-diabetic subjects. PLoS One. 2020 Oct 7;15(10):e0237733. doi: 10.1371/journal.pone.0237733. eCollection 2020. PMID 33027294
- [Background] Hanewinckel R, van Oijen M, Taams NE, Merkies ISJ, Notermans NC, Vrancken AFJE, Ikram MA, van Doorn PA. Diagnostic value of symptoms in chronic polyneuropathy: The Erasmus Polyneuropathy Symptom Score. J Peripher Nerv Syst. 2019 Sep;24(3):235-241. doi: 10.1111/jns.12328. Epub 2019 Jul 9. PMID 31172622
- [Background] Hanewinckel R, Drenthen J, van Oijen M, Hofman A, van Doorn PA, Ikram MA. Prevalence of polyneuropathy in the general middle-aged and elderly population. Neurology. 2016 Nov 1;87(18):1892-1898. doi: 10.1212/WNL.0000000000003293. Epub 2016 Sep 28. PMID 27683845
- [Background] Ferdousi M, Azmi S, Kalteniece A, Khan SU, Petropoulos IN, Ponirakis G, Alam U, Asghar O, Marshall A, Soran H, Boulton AJM, Augustine T, Malik RA. No evidence of improvement in neuropathy after renal transplantation in patients with end stage kidney disease. J Peripher Nerv Syst. 2021 Sep;26(3):269-275. doi: 10.1111/jns.12456. Epub 2021 Jun 10. PMID 34085731
- [Derived] Nolte S, Shehab NBN, Berger SP, Oldag C, Nolte IM, de Greef BTA, Lange F, van Londen M, Faber CG, Bakker SJL, van Doorn PA, Moes HR, Drost G. Polyneuropathy in Kidney Transplant Recipients: Accuracy of a New Clinical Diagnostic Scoring System. J Peripher Nerv Syst. 2025 Sep;30(3):e70058. doi: 10.1111/jns.70058. PMID 40915314